CLINICAL TRIAL: NCT00088088
Title: A Phase I/II Trial of STA-4783 in Combination With Paclitaxel and Carboplatin for the Treatment of Chemotherapy Naive Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: STA-4783 in Combination With Paclitaxel and Carboplatin for the Treatment of Chemotherapy Naive Patients With Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4783-02
Record Dates: First submitted 2004-07-20; First posted 2004-07-21 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; elesclomol

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin
Drug: STA 4783

SUMMARY:
This study is for patients who have Stage IIIb or Stage IV NSCLC and have never had chemotherapy before for their disease. The first phase of the study recently completed and for the second phase of the study patients are randomly assigned to receive either paclitaxel and carboplatin or paclitaxel and carboplatin and study drug (STA 4783). Treatment will be every 3 weeks for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven NSCLC (mixed forms with small cell lung cancer are excluded) with clinically stage IIIB or stage IV disease.
* No prior systemic chemotherapy treatment.
* Prior treatments with radiotherapy or local ablative therapies are allowed if these therapies do not affect the measurable target lesions being used for the purposes of this protocol. Completion of any radiotherapy must be greater than or equal to 4 weeks prior to study entry, and/or resolution of all acute toxic effects of any prior radiotherapy or major surgical procedure to National Cancer Institute (NCI) Common Toxicity Criteria (CTC) grade less than or equal to 1.
* Evidence of unidimensionally measurable disease (ie, greater than or equal to 1 malignant tumor mass that may be accurately measured in at least 1 dimension greater than or equal to 20 mm with conventional radiographic techniques or magnetic resonance imaging [MRI], or greater than or equal to 10 mm with spiral computerized tomography [CT] scan). Tumor evaluation by positron emission tomography (PET) scan or by ultrasound may not substitute for CT or MRI scans. Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions, and disease documented by indirect evidence only (eg, by laboratory tests such as alkaline phosphatase) are not considered measurable.
* Female or male, 18 years of age or older.
* ECOG performance status 0 or 1.
* Neuropathy of Grade 0 or Grade 1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate aminotransferase (AST; serum glutamate-oxalate transferase [SGOT]) and serum alanine aminotransferase (ALT; serum glutamate-pyruvate transferase) [SGPT] less than or equal to 2.5 x central laboratory upper limit of normal (ULN). If liver function abnormalities are due to underlying malignancy, then AST and ALT may be less than or equal to 5 x ULN.
  * Total serum bilirubin less than or equal to 1.5 x ULN
  * Prothrombin time (PT) and partial thromboplastin time (PTT) less than or equal to 1.5x ULN
  * Absolute neutrophil count (ANC) greater than or equal to 1500/mL
  * Platelets greater than or equal to 100,000/mL
  * Hemoglobin greater than or equal to 9.0 g/dL
  * Serum creatinine less than or equal to 1.5 x ULN
* The effects of STA-4783 on the developing human fetus are unknown, however, taxanes and platinum analogues are known to be teratogenic. Therefore, women of childbearing potential (defined as, unless surgically sterile, women <=50 years of age or history of amenorrhea for < 12 months prior to study entry) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she must agree to inform the treating physician immediately, and be followed until delivery.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Patients with large untreated pleural effusions, or who have immediate life-threatening complications of their disease, or those who may need urgent radiotherapy (e.g., due to lobar obstruction, painful bony sites, cord compression, or superior vena cava syndrome).
* Current participation in another clinical drug trial; may not be receiving an investigational drug or any other agent that has an immunomodulatory or presumed anti-tumor effect within 4 weeks of study entry.
* Known brain metastases, or leptomeningeal disease on screening CT or MRI scan, except for treated disease that is considered clinically and radiologically stable, and does not require treatment with anti-convulsants and/or steroids.
* Prior malignancy other than NSCLC within the last 5 years with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal or squamous cell carcinoma of the skin;
  * Previous nonpulmonary malignancy confined and surgically resected with no evidence of active malignancy.
* Has a known allergy to Cremophor® or Cremophor®-based drug products.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Pregnancy or breast feeding.
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2004-03; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - NEA Clinic, Jonesboro, Arkansas
  - Wilshire Oncology Medical Group, Pomona, California
  - St. Francis Memorial Hospital, San Francisco, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Kaiser Permanete, Vallejo, California
  - Oncology Associates of Bridgeport, Trumball, Connecticut
  - ACORN, Miami, Florida
  - Oncology Hematology Consultants, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - The Cancer Institute at Alexian Brothers, Elk Grove Village, Illinois
  - Ingalls Hospital, Harvey, Illinois
  - Overton Brooks, VAMC, Shreveport, Louisiana
  - LSUHSC - Shreveport Feist Weiller Cancer Center, Shreveport, Louisiana
  - Maryland Hematology and Oncology Associates, Baltimore, Maryland
  - The Duluth Clinic, Duluth, Minnesota
  - The West Clinic, Memphis, Tennessee
  - The Sarah Cannon Research Center, Nashville, Tennessee
  - Presbyterian Hospital, Dallas, Texas
  - Multicare Health System, Tacoma, Washington